CLINICAL TRIAL: NCT03465345
Title: Phase 1b Study of Metformin Plus Oligomeric Procyanidin Complex for Pharmacologic Manipulation of AGE (Advanced Glycation Endproducts) Levels in Prostate Cancer Patients
Brief Title: Study of Metformin Plus Oligomeric Procyanidin Complex for Pharmacologic Manipulation of AGE (Advanced Glycation Endproducts) Levels in Prostate Cancer Patients
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was stopped to pursue a new treatment plan with a new study.
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 102797
Record Dates: First submitted 2018-02-27; First posted 2018-03-14 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Metformin + OPC dose escalation (Experimental)
  Interventions: Drug: Metformin; Drug: Oligomeric Procyanidin Complex

INTERVENTIONS:
Drug: Metformin — Metformin: The starting dose for Metformin is 850mg once a day, the second dose is 850mg once a day; the third dose level is 850mg twice a day; the fourth dose level is 850mg twice a day. Each dose level lasts for 28 days.
Drug: Oligomeric Procyanidin Complex — OPC: The starting dose for OPC is 500mg once a day; the second dose is 1000mg once a day; the third dose level is 1000mg once a day; the fourth dose level is 1500mg once a day. Each dose level lasts for 28 days.
  Other Names: OPC

SUMMARY:
The overall goal of this study is to identify a safe dose of metformin, in combination with oligomeric procyanidin complex (OPC) for pharmacologic reduction of AGE levels in patients with prostate cancer.

DETAILED DESCRIPTION:
AGEs (advanced glycation endpoints) are a type of metabolite, or substance, found in the food. The AGE content in food is determined by the types of food you eat and also how you prepare your food. The researchers helping conduct this study have found a potential link between AGE levels and cancer. The purpose of this study is to identify safe pharmaceutical agents that can reduce the AGE levels in subjects with advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmation of adenocarcinoma of the prostate that is documented by one of the following: pathology report or clinic note with documented history of prostate cancer.
2. Subjects must be receiving ADT with a GnRH agonist or antagonist, with or without an anti-androgen, with a current testosterone level documented to be <50ng/dL at enrollment. Subjects whose ADT is interrupted may enroll or continue on study as long as the testosterone is documented to remain <50ng/dL for the entire duration of study participation. Subjects who have undergone orchiectomy are also eligible.
3. Subjects must have adequate hematologic, renal, and hepatic function at baseline, as follows:

   * Hematology parameters: ANC >1000/mcL, platelets > 100,000/mcL, Hgb >8.0gm/dL
   * Renal Function: eGFR of ≥ 45mls/min using Cockkroft and Gault formula (see appendix C).
   * Liver Function: Total bilirubin ≤ULN, AST and ALT <1.5xULN, Prior radiation therapy allowed
4. Subjects may have diabetes mellitus but must not be taking metformin.
5. Able to swallow and retain oral medication
6. ECOG performance status of 0 - 2
7. Ability to sign written informed consent
8. Testosterone level <50ng/dL at time of enrollment.
9. Age 18 or older.

Exclusion Criteria:

1. Known allergy to grapes or grape seed
2. Known hypersensitivity or intolerance to metformin.
3. Any condition associated with increased risk of metformin-associated lactic acidosis (e.g. congestive heart failure defined as NYHA Class III or IV functional status, history of acidosis of any type; habitual intake of 3 or more alcoholic beverages per day).
4. Prior cytotoxic chemotherapy for metastatic prostate cancer; prior treatment with genomically-targeted agents, or Provenge is allowed.
5. History of receiving more than 2 classes of ADT.
6. Current use of metformin, or strong antioxidants (extracts from grape seed, milk thistle; pine bark, green tea, saw palmetto; resveratrol; flavonoids; catechins; ellagic acid), large quantities of red grapes, white button mushrooms, red wine
7. PSA doubling time of <6 months, measured over the 3 months prior to enrollment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2018-07-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of metformin in combination with OPC in PCa subjects. | 112 days

SECONDARY OUTCOMES:
Correlation between changes to AGE level and changes to PSA. | 112 days
Correlation between changes to AGE level and changes to BMI. | 112 days
Correlation between changes to AGE level and changes to insulin resistance. | 112 days
Correlation between changes to AGE level and changes to A1C. | 112 days
Correlations between changes to AGE level and changes to testosterone. | 112 days
Correlation between changes to AGE level and changes to diet. | 112 days
Correlation between changes to AGE level and changes to quality of life. | 112 days
  FACT-P and AUA questionnaires
Frequency of adverse events as assessed by CTCAE v. 4 | 112 days
  Toxicities will be tabulated by type and grade and the proportion of patients with grade 3, grade 4 or an SAE will be estimated with a 90% confidence interval.
Correlation between AGE levels and sRAGE (soluble receptor for AGE) expression and signaling. | 112 days
Correlation between changes to AGE level and OPC metabolite levels. | 112 days
Correlation between changes to AGE level and changes in the stool. microbiome. | 112 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lilly, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No